CLINICAL TRIAL: NCT01746173
Title: A Phase II Study of CHOEP Induction Followed by Gemcitabine/Busulfan/Melphalan Autologous Stem Cell Transplantation for Patients With Newly Diagnosed T-Cell Lymphoma
Brief Title: CHOEP + High Dose Therapy + Auto SCT for T-Cell Lymphoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual and futility
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Massachusetts General Hospital (Other); Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Philippe Armand, MD, PhD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-388
Record Dates: First submitted 2012-12-04; First posted 2012-12-10 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: T-cell Non-Hodgkin Lymphoma
Keywords: T Cell lymphoma
MeSH Terms: conditions — Lymphoma, T-Cell | interventions — Cyclophosphamide; Doxorubicin; Vincristine; Etoposide; etoposide phosphate; Prednisone; Filgrastim; Granulocyte Colony-Stimulating Factor; plerixafor; Leukapheresis; Fibroblast Growth Factor 7; Gemcitabine; Busulfan; Melphalan; Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CHOEP + High Dose Therapy + Auto SCT (Experimental): Patients received 6 cycles of induction chemotherapy: Cyclophosphamide, Doxorubicin, Vincristine, Etoposide and Prednisone (CHOEP) (5 if previously received 1 cycle of CHOP). CHOP was given at standard doses, with a dose of etoposide of 100 mg/m2 intravenously (IV) or 200 mg/m2 orally added on days 1-3 of each cycle. Patients who did not achieve a partial (PR) or complete (CR) remission at restaging after either 3 or 6 cycles were taken off study. Responders after 6 cycles had stem cell (SC) mobilization using filgrastim and plerixafor (if necessary) within 4 weeks of the end of induction. SC mobilization, harvesting, and reinfusion were performed per standard institutional protocol. A minimum collection of 2x106 CD34+ cells/kg was required to proceed to autologous stem cell transplant. Conditioning was comprised of gemcitabine 2700 mg/m2 on days -8 and -3, IV busulfan 105 mg/m2 days -8 to -5, and melphalan 60 mg/m2 given daily on days -3 and -2 (per MD Andersen protocol).
  Interventions: Drug: Cyclophosphamide; Drug: Doxorubicin; Drug: Vincristine; Drug: Etoposide; Drug: Prednisone; Drug: Filgrastim; Drug: Plerixafor; Procedure: Stem Cell Collection; Drug: Palifermin; Drug: Gemcitabine; Drug: Busulfan; Drug: Melphalan; Procedure: Stem Cell Transplant

INTERVENTIONS:
Drug: Cyclophosphamide
  Other Names: cytoxan
Drug: Doxorubicin
  Other Names: adriamycin
Drug: Vincristine
  Other Names: oncovin
Drug: Etoposide
  Other Names: Etopophos; Toposar; Etoposide phosphate
Drug: Prednisone
Drug: Filgrastim
  Other Names: neupogen; G-CSF
Drug: Plerixafor
  Other Names: mozobil
Procedure: Stem Cell Collection
  Other Names: Leukapheresis
Drug: Palifermin
  Other Names: KGF; kepivance
Drug: Gemcitabine
  Other Names: gemzar
Drug: Busulfan
  Other Names: busulfex
Drug: Melphalan
Procedure: Stem Cell Transplant
  Other Names: Stem Cell Infusion

SUMMARY:
The current standard of care for the frontline treatment of peripheral T-cell lymphomas (PTCL) is induction chemotherapy followed by autologous stem cell transplantation (ASCT). However, many patients are unable to get to ASCT or relapse after ASCT, with a poor prognosis. Recently, a novel ASCT conditioning regimen of gemcitabine, busulfan and melphalan (Gem/Bu/Mel) has been reported to lead to favorable outcomes in this disease. We therefore designed a frontline regimen of CHOEP induction followed by Gem/Bu/Mel ASCT, and report the results of a phase 2 study of this regimen in patients with PTCL.

DETAILED DESCRIPTION:
Objectives:

Primary

* To estimate the proportion of patients alive and progression-free at 24 months after beginning induction therapy

Secondary

* To estimate the response rate (complete remission (CR) and partial remission (PR)) after CHOEP x 6 and after Gem/Bu/Mel ASCT
* To estimate overall survival (OS), progression-free survival (PFS), cumulative incidence of relapse (CIR), and non-relapse mortality (NRM)
* To estimate the toxicity (grade 3 and above)
* To estimate the rate of successful stem cell mobilization after CHOEP in responding patients
* To estimate the proportion of patients who can successfully complete the entire treatment regimen
* To estimate the time to engraftment of neutrophil and platelet engraftment after ASCT
* To determine whether tumor DNA can be detected in peripheral blood of patients before therapy
* To evaluate the changes and prognostic relevance in detectable tumor DNA in peripheral blood after induction chemotherapy (CHOEP) and after Gem/Bu/Mel ASCT

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of T-Cell lymphoma with mandatory pathologic review at Brigham and Women's Hospital or Massachusetts General Hospital
* Measurable disease
* Candidate for Autologous Stem Cell Transplant

Exclusion Criteria:

* Prior anti-lymphoma chemotherapy (except steroids/radiotherapy for urgent palliation, one prior cycle of CHOP or up to 2 prior cycles of CHOEP)
* Pregnant or breastfeeding
* Alk-positive ACL
* Significant neuropathy precluding vincristine administration
* Known hypersensitivity to any of the agents used in the treatment
* Uncontrolled intercurrent illness
* Receiving other investigational agents
* History of a different malignancy except if disease free for at least 5 years or have cervical cancer in situ or basal cell/squamous cell carcinoma of the skin
* HIV positive on anti-retroviral therapy

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Armand, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 patients were enrolled between July 2013 and January 2014.
Period: Overall Study
Arm/Group | CHOEP + High Dose Therapy + Auto SCT
Started | 5
Completed | 3
Not Completed | 2
Not completed — Disease Progression | 2

BASELINE CHARACTERISTICS:
Population: The analysis dataset is comprised of all enrolled patients.
Arm/Group | CHOEP + High Dose Therapy + Auto SCT
Number analyzed (Participants) | 5
Age, Continuous [Mean (Full Range); unit: years] | 55 [39 to 69]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5
Stage [Count of Participants; unit: Participants] — Stage per Ann Arbor Classification
  Participants
    Stage I | 1
    Stage II | 0
    Stage III | 2
    Stage IV | 2

OUTCOME MEASURES:

1. Primary Outcome: 24-month Progression-Free Survival Rate
Description: 24-month progression-free survival rate is defined as the proportion of patients remaining alive and progression-free at 24 months from start of induction therapy. Disease progression was assessed using a combination of CT scans and PET scans. Progression was categorized according to standard lymphoma response criteria, specifically the Revised Response Criteria (Cheson 2007).
Time Frame: Disease was re-staged at cycles 3 and 6 during induction, at day 100 post-ASCT, and in long-term follow-up at months 12, 18, 24 and 36. All patients were evaluable up to month 24.
Population: The analysis dataset is comprised all enrolled patients.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | CHOEP + High Dose Therapy + Auto SCT
Number analyzed (Participants) | 5
proportion of patients | 0.0 [0.0 to 0.45]

2. Secondary Outcome: Induction Response
Description: Induction response is the defined as the proportion of patients who achieve complete remission (CR) or partial remission (PR) during 6 cycles of induction therapy. Response was assessed was using a combination of CT scans and PET scans. Partial and complete response were categorized according to standard lymphoma response criteria, specifically the Revised Response Criteria (Cheson 2007). Given the cycle length of 3 weeks, induction duration per protocol was 18 weeks.
Time Frame: Disease was re-staged at cycles 3 and 6 during induction. Median duration of induction therapy in this study cohort was 6 cycles/18 weeks (range 2-6 cycles).
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | CHOEP + High Dose Therapy + Auto SCT
Number analyzed (Participants) | 5
proportion of patients | .60 [.19 to .92]

ADVERSE EVENTS:
Time Frame: Toxicity was assessed weekly during 6 cycles of induction (up to 18 weeks), within 0-3 days prior to day 1 of stem cell mobilization, day +30 post-ASCT. Median duration of induction therapy was 6 cycles/18 weeks (range 2-6 cycles). 3 patients continued to ASCT within 7 months of study enrollment.
Description: Maximum grade toxicity by type was first calculated. Serious AEs were defined as events with treatment attribution of possibly, probably or definitely and grade 3 or higher per CTCAEv4. Other AEs were defined as events with treatment attribution of possible, probable or definite and grades 1 or 2 per CTCAEv4. No further data is available to specify classification of other beyond the general term.
Arm/Group | CHOEP + High Dose Therapy + Auto SCT
Serious Adverse Events (participants affected / at risk) | 4/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHOEP + High Dose Therapy + Auto SCT (N=5)
Anemia (Blood and lymphatic system disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 2
Platelet count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CHOEP + High Dose Therapy + Auto SCT (N=5)
Anemia (Blood and lymphatic system disorders) | 1
Anal stenosis (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Chills (General disorders) | 1
Edema limbs (General disorders) | 1
Fatigue (General disorders) | 3
Fever (General disorders) | 1
Infections and infestations - Other (Infections and infestations) | 1
Neutrophil count decreased (Investigations) | 1
White blood cell decreased (Investigations) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
The trial closed early due to poor accrual. The small sample size precludes definitive conclusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No